CLINICAL TRIAL: NCT04560569
Title: A Multicenter, Two-Arm, 24-Week Study of Albuvirtide in Combination With 3BNC117 in Patients With Multi-Drug Resistant (MDR) HIV-1 Infection
Brief Title: Albuvirtide in Combination With 3BNC117 in Patients With Multi-Drug Resistant (MDR) HIV-1 Infection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Frontier Biotechnologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABT-3BNC117_203
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-01

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — albuvirtide; 3BNC117 antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): ABT weekly and 3BNC117 bi-weekly
  Interventions: Drug: Albuvirtide; Drug: 3BNC117 Antibody
- Group B (Experimental): both ABT and 3BNC117 treatment bi-weekly
  Interventions: Drug: Albuvirtide; Drug: 3BNC117 Antibody

INTERVENTIONS:
Drug: Albuvirtide — Long-Acting HIV-1 Fusion Inhibitor (chemically modified peptide targeting HIV-1 gp41)
  Other Names: ABT
Drug: 3BNC117 Antibody — Recombinant, fully human mAb of the IgG1κ isotype that specifically binds to HIV-1 gp120
  Other Names: 3BNC117

SUMMARY:
The primary objectives are to assess the antiviral activity, clinical safety and tolerability parameters of albuvirtide/3BNC117 combination therapy in reducing HIV-1 viral load during the 1-week induction period treatment period.

DETAILED DESCRIPTION:
This is a Phase 2, multi-center study to evaluate the efficacy, safety, and tolerability of ABT/3BNC117 combination in conjunction with an existing failing antiretroviral therapy (ART) for 1 week, and then with optimized background regimen (OBR) for 24 weeks, respectively. A total of 20 eligible subjects who demonstrate evidence of HIV-1 replication despite ongoing antiretroviral therapy with documented genotypic and/or phenotypic resistance to multiple classes of HIV drugs (3 classes or more) will be enrolled. Patients must have been treated with HAART for at least 6 months and be failing or have recently failed (i.e., in the last 8 weeks) therapy to determine baseline viral load.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, age ≥ 18 years;
2. HIV-1 seropositive with documented HIV-1 infection by official, signed, written history (e.g. Laboratory report)
3. Receiving a combination antiretroviral therapy (cART) (failing regimen) for at least 8 weeks before Screening and are willing to continue on the failing regimen during the Screening Phase and up to Day 14 of the Treatment Phase, OR have failed in the past 8 weeks of Screening, are off therapy and are willing to stay off therapy until Day 14 of the Treatment Phase;
4. Plasma HIV-1 RNA ≥ 1000 copies/mL at the Screening Visit and documented detectable viral load (HIV-1 RNA >200 copies/ml) within the last 3 months prior to the Screening Visit;
5. Highly treatment-experienced HIV-infected patients with genotypic and/or phenotypic resistance to at least one ARV drug for each of three or more drug classes of antiretroviral medications at the Screening Visit and have difficulty in constructing a viable suppressive regimen;
6. Have full viral sensitivity/susceptibility to at least one approved antiretroviral agent, other than ABT and 3BNC117, as determined by genotypic and/or phenotypic ARV drug resistance tests at screening, and such agent can be used as a component of OBR;
7. Be willing to remain on treatment without any changes or additions to the OBR regimen, except for toxicity management or upon meeting criteria for treatment failure;
8. Have a life expectancy that is > 9 months;
9. Laboratory values at Screening of:

   1. Absolute neutrophil count (ANC) ≥ 750/mm3;
   2. Hemoglobin (Hb) ≥ 10.5 gm/dL (male) or ≥ 9.5 gm/dL (female);
   3. Platelets ≥ 75,000 /mm3;
   4. Serum alanine transaminase (SGPT/ALT) < 1.25 x upper limit of normal (ULN);
   5. Serum aspartate transaminase (SGOT/AST) < 1.25 x ULN;
   6. Serum total bilirubin within normal range; and
   7. Creatinine ≤ 1.5 x ULN.
10. Clinically normal resting 12-lead electrocardiogram (ECG) at the Screening Visit or, if abnormal, considered not clinically significant by the Principal Investigator
11. Both male and female patients and their partners of childbearing potential must agree to use 2 medically accepted methods of contraception (e.g., barrier contraceptives [male condom, female condom, or diaphragm with a spermicidal gel], hormonal contraceptives [implants, injectables, combination oral contraceptives, transdermal patches, or contraceptive rings], and intrauterine devices) during the course of the study (excluding women who are not of childbearing potential and men who have been sterilized). Females of childbearing potential must have a negative serum pregnancy test at the Screening visit and negative urine pregnancy test prior to receiving the first dose of study drug; and
12. Willing and able to participate in all aspects of the study, including use of IV medication, completion of subjective evaluations, attendance at scheduled clinic visits, and compliance with all protocol requirements as evidenced by providing written informed consent.

Note: Subjects diagnosed with either substance dependence or substance abuse or any history of a concomitant condition (e.g., medical, psychological, or psychiatric) may be enrolled if, in the opinion of site investigator these circumstances would not interfere with the subject's successful completion of the study requirements.

Exclusion Criteria:

1. Subject having ≥0.5 log10 reduction in HIV-1 RNA viral load from the Screening Visit to Baseline Visit (Day 0).

   Note: This criterion will be evaluated prior to randomization at T1 Visit (Day 7).
2. Any active infection or malignancy requiring acute therapy;
3. Hepatitis B infection as manifest by the presence of Hepatitis B surface antigen (HBsAg);
4. Hepatitis C infection as manifest by positive anti-HCV antibody and positive HCV RNA assay at the time of screening;
5. Grade 4 DAIDS laboratory abnormality;
6. Females who are pregnant, lactating, or breastfeeding, or who plan to become pregnant during the study;
7. Unexplained fever or clinically significant illness within 1 week prior to the first study dose;
8. Any vaccination within 2 weeks prior to the first study dose;
9. Prior exposure to albuvirtide or 3BNC117
10. Subjects weighing <35kg;
11. History of anaphylaxis to any oral or parenteral drugs;
12. Use of any fusion inhibitors (T20) and broadly neutralizing monoclonal antibody prior to the Screening Visit, including the investigational drugs, or having documented genotypic and/or phenotypic resistance to fusion inhibitors;
13. Participation in an experimental drug trial(s) within 30 days of the Screening Visit;
14. Any known allergy or antibodies to the study drug or excipients;
15. Treatment with any of the following:

    1. Radiation or cytotoxic chemotherapy with 30 days prior to the screening visit;
    2. Immunosuppressants or immunomodulating agents within 60 days prior to the screening visit; or
    3. Oral or parenteral corticosteroids within 30 days prior to the Screening Visit. Subjects on chronic steroid therapy 5 mg/day will be excluded with the following exception:

       * Subjects on inhaled, nasal, or topical steroids will not be excluded.
16. Any other clinical condition that, in the Investigator's judgment, would potentially compromise study compliance or the ability to evaluate safety/efficacy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-30 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with ≥0.5 log10 reduction in HIV-1 RNA viral load from baseline (Day 7) to Day 14 as compared to the control period from Day 0 to Day 7. | Day 14
  Proportion of participants (%) achieving a viral load reduction of at least 0.5 log from baseline (Day 7)

SECONDARY OUTCOMES:
Mean change in HIV-1 RNA levels (log10 copies/mL) from baseline (Day 7) to Day 14 as compared to the control period from Day 0 to Day 7. | Day 14
  Mean change in HIV-1 RNA levels from Day 7 to Day 14
Mean change in CD4+/CD8+ T cell count from baseline (Day 7) to Day 14 as compared to the control period from Day 0 to Day 7. | Day 14
  Mean change in CD4+/CD8+ T cell count from Day 7 to Day 14
Percentage of participants achieving HIV-1 RNA <200 copies/mL at the EOT. | Week 25/EOT
  Percentage of participants achieving HIV-1 RNA <200 copies/mL
Mean change in HIV-1 RNA levels (log10 copies/mL) during the course of Treatment Phase | Through Week 25/EOT
  Mean change in HIV-1 RNA levels from Day 0 to EOT
Mean change in HIV-1 RNA levels (log10 copies/mL) from baseline (Day 7) to EOT. | Week 25/EOT
  Mean change in HIV-1 RNA levels from Day 7 to EOT
Mean change in CD4+/CD8+ T cell count from baseline (Day 7) to EOT. | Week 25/EOT
  Mean change in CD4+/CD8+ T cell count from Day 7 to EOT

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Yao, M.D., Study Director — Frontier Biotechnologies Inc.
Locations (7):
- United States (7):
  - ABT-3BNC117_203 Investigational Site, Canoga Park, California
  - ABT-3BNC117_203 Investigational Site, San Francisco, California
  - ABT-3BNC117_203 Investigational Site, Hialeah, Florida
  - ABT-3BNC117_203 Investigational Site, Orlando, Florida
  - ABT-3BNC117_203 Investigational Site, West Palm Beach, Florida
  - ABT-3BNC117_203 Investigational Site, Decatur, Georgia
  - ABT-3BNC117_203 Investigational Site, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No